CLINICAL TRIAL: NCT04823559
Title: The ThinkCancer! Intervention: Protocol for a Feasibility Study Incorporating a Randomised Pilot Trial With an Embedded Process and Economic Evaluation
Brief Title: The ThinkCancer! Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangor University (Other)
Collaborators: Cancer Research Wales (Unknown); North Wales Organisation for Randomised Trials in Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UWalesBangor
Record Dates: First submitted 2020-12-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual practice (No Intervention): Usual practice
- Intervention (Experimental): Receives educational workshop
  Interventions: Other: ThinkCancer workshop

INTERVENTIONS:
Other: ThinkCancer workshop — The proposed intervention, the ThinkCancer! Workshop, is practice-based and consists of themed sessions for both clinical and non-clinical staff, the co-production of a Cancer Safety Netting Plan (CSNP) and the appointment of a Cancer Safety Netting Champion (CSNC). The workshop aims to raise awareness and increase knowledge around current cancer diagnosis guidance and will be delivered over half a day during GP protected time in the form of face-to-face educational sessions. Sessions will consist of a series of interactive activities exploring existing processes within practices and developing plans for change to implement each component.
  Arms: Intervention

SUMMARY:
Background Wales, like other UK countries, has relatively poor cancer outcomes. Late diagnosis and a slow referral process are major contributors. General practitioners (GPs) and other care providers working in primary care are often faced with patients presenting with a multitude of non-specific symptoms that could be cancer. Safety netting can be used to manage diagnostic uncertainty by ensuring patients with vague symptoms are appropriately monitored. The ThinkCancer! Workshop is an educational behaviour change intervention aimed at the whole general medical practice team, designed to improve primary care approaches to ensure timely diagnosis of cancer. The workshop will consist of teaching and awareness sessions, appointment of a Safety Netting Champion and the development of a bespoke Safety Netting Plan. This study aims to assess the feasibility of the ThinkCancer! Intervention for a future definitive randomised controlled trial, in terms of recruitment, randomisation, retention, acceptability, adherence and barriers to the intervention.

Methods The ThinkCancer! study is a randomised, multisite feasibility trial, with an embedded process evaluation and economic evaluation. Twenty-three to 30 general medical practices will be recruited across Wales, randomised in a ratio of 2:1 of intervention versus control who will follow usual care. The workshop will be delivered by a GP educator, and will be adapted iteratively throughout the trial period. Baseline practice characteristics will be collected via questionnaire. We will also collect Primary Care Interval (PCI), Two Week Wait (2WW) referral rate, conversion rate and detection rate at baseline and six months post-randomisation. Participant feedback, researcher reflective notes and economic costings will be collected following each workshop. A process evaluation will assess implementation using an adapted Normalisation Measure Development (NoMAD) questionnaire and qualitative interviews. An economic feasibility analysis will inform a future economic evaluation.

Discussion This study will allow us to test and further develop a novel evidenced-based complex intervention aimed at general practice teams to expedite the diagnosis of cancer in primary care. The results from this feasibility study will inform the future design of a full-scale definitive phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Any practices in Wales are eligible for inclusion.

Exclusion Criteria:

* As we intend to include a broad group of general medical practices, there are no formal exclusion criteria.

As determining feasibility is the main objective of this study, the eligibility criteria remain broad in order to allow for inclusion of a range of practices, which will aid the intervention refinement and allow for a better understanding on what is feasible in all types of practices and why some practices may not take part.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a future definitive trial | From date of initial expression of interest to participate to end of follow up period (13 months)
  Number of practices approached, interested in participating, consented and randomised, retention of recruited practices, ability to collect data

SECONDARY OUTCOMES:
Two Week Wait referral rate | Six months pre-randomisation and six months post-randomisation
  Number of two week rate referrals made in a given time period, multiplied by 100000 and divided by the practice list size
Primary Care Interval | Six months pre-randomisation and six months post-randomisation
  The time between the date of first presentation and the date of referral

CONTACTS AND LOCATIONS:
Overall Officials: Clare Wilkinson, Principal Investigator — Bangor University
Locations (7):
- United Kingdom (7):
  - Betsi Cadwaldr University Health Board, Bangor
  - Aneurin Bevan University Health Board, Blaenau Gwent
  - Hywel Dda University Health Board, Camarthenshire
  - Cardiff and Vale University Health Board, Cardiff
  - Cwm Taf Morgannwg University Health Board, Cwm Taf
  - Powys Teaching Health Board, Powys
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Disbeschl S, Surgey A, Roberts JL, Hendry A, Lewis R, Goulden N, Hoare Z, Williams N, Anthony BF, Edwards RT, Law RJ, Hiscock J, Carson-Stevens A, Neal RD, Wilkinson C. Protocol for a feasibility study incorporating a randomised pilot trial with an embedded process evaluation and feasibility economic analysis of ThinkCancer!: a primary care intervention to expedite cancer diagnosis in Wales. Pilot Feasibility Stud. 2021 Apr 21;7(1):100. doi: 10.1186/s40814-021-00834-y. PMID 33883033